CLINICAL TRIAL: NCT05927259
Title: The Role of N-acetylcysteine as a Novel Adjuvant Treatment in Acute Organophosphorus.A Randomized, Clinical Trial in Poison Control Center -Ain Shams University Hospitals
Brief Title: The Role of N-acetylcysteine as a Novel Adjuvant Treatment in Acute Organophosphorus Pesticide Poisoning
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Saeed Mohammed, lecturer of clinical toxicology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R214/2021
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Acute Organophosphorus Poisoned Patients
MeSH Terms: interventions — Acetylcysteine; Atropine; Oximes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Patients who will receive (conventional treatment of acute organophosphorus poisoning plus NAC)
  Interventions: Drug: n acetyl cysteine; Drug: standard treatment
- control group (Other): Patients who will receive conventional treatment only
  Interventions: Drug: standard treatment

INTERVENTIONS:
Drug: n acetyl cysteine — A patients received NAC 140 mg/Kg IV infusion (as a loading dose), then 70 mg/KgIV infusion every 4 hours up to 17 doses
  Arms: study group
Drug: standard treatment — stabilization and antidotes
  Other Names: atropine and oximes

SUMMARY:
All patients admitted in the ICU of the PCC-ASUH due to acute poisoning by acute organophosphorus poisoning will be included in the study. The diagnosis of intoxication will be based on history of acute exposure , clinical examination and laboratory investigations. Patients will be randomly allocated into 2 equal groups.

Group 1 -. Patients who will receive (conventional treatment of acute organophosphorus poisoning plus NAC) and Group 2 - Patients who will receive conventional treatment only

DETAILED DESCRIPTION:
40 patients with acute organophosphorus poisoning will be randomly assigned as control groups and study group in a 1:1 ratio ( 20 patients in each group). The diagnosis of acute organophosphorus intoxication will be based on history of acute exposure, clinical examination and laboratory investigations. Patients will be randomly allocated into 2 equal groups.

Group 1 - Patients who will receive (conventional treatment of acute organophosphorus poisoning plus NAC) Group 2 - Patients who will receive conventional treatment only

ELIGIBILITY:
Inclusion Criteria:

All patients (above 16 years) admitted to the ICU of the PCC-ASUH due to acute poisoning by acute organophosphorus poisoning will be included in the study. The diagnosis of intoxication will be based on history of acute exposure, clinical examination and laboratory investigations. -

Exclusion Criteria:

* Based on the possibility of alteration in measured parameters and/or biomarkers, patients below 16 years or above 60 years Patients with history of diabetes, cardiac disease, respiratory, renal disease and hepatic disease.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
mortality | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sarah S Mohammed, Principal Investigator — faculty of medicine ain shams university
Locations (3):
- Egypt (3):
  - faculty of medicine Ain shams university, Cairo, None Selected
  - Faculty of Medicine, Cairo, None Selected
  - Poison Control Center Ain Shams University Hospitals, Cairo

IPD SHARING:
Plan to Share IPD: No